CLINICAL TRIAL: NCT03790397
Title: A Retrospective, Multicenter and Observational Study of Osimertinib Monotherapy Treatment in Subjects With Advanced or Metastatic Non-Small Cell Lung Cancer EGFR-T790M Mutation-positive Who Have Received the Treatment Within the Special Use Medication Program in Spain
Brief Title: Osimertinib in Subjects With Advanced Non-Small Cell Lung Cancer EGFR-T790M Mutation-positive
Acronym: OSIREX
Status: Completed | Type: Observational
Sponsor: Fundación GECP (Other)
Responsible Party: Sponsor
Other Study IDs: GECP 18/01_OSIREX
Record Dates: First submitted 2018-12-24; First posted 2018-12-31 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Lung Cancer, EGFR positive, NSCLC, Osimertinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — osimertinib; atezolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Osimertinib — Patients treated with Osimertinib within the Special Use medication Program (SUMP).
  Other Names: Tecentriq

SUMMARY:
This is a retrospective, multicenter and observational study of Osimertinib monotherapy treatment in Subjects with advanced or metastatic Non-Small Cell Lung Cancer (NSCLC) EGFR-T790M mutation-positive who have received the treatment within the Special Use Medication Program (SUMP) in Spain.

DETAILED DESCRIPTION:
The study is based on the collection of data about the patients treated with Osimertinib within the Special Use medication Program. the patienes participating in this non-interventional study will not receive treatment in relation to the study.

Approximately a total of 270 patients will be included in this project from several Spanish sites. Around 52 hospitals will participate in the study. the observation period is from August 2016 to December 2018 and will include patients who started the treatment with Osimertininb from August 2016 to April 2018.

The primary objective is to estimate the progression free survival of the Osimertinib treatment.

ELIGIBILITY:
Inclusion Criteria:

* Squamous or Non-Squamous, non-small cell lung cancer (NSCLC), Stage IIIb/IV (histologically or cytologically confirmed), EGFRm/T790M, who received osimertinib treatment within the Spanish special use medication program of Osimertinib (SUMP).
* Alive patients must have signed, dated and IRB/EC-approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol-related procedures that are not part of normal subject care.

Exclusion Criteria:

* Alive patients who do not want to sign and date an IRB/IEC-approved written informed consent form.
* Patients who were accepted in the SUMP, but did not receive treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who have received Osimertinib in the SUMP in Spain.
Sampling Method: Non-Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Progression free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  To estimate the progression free survival of the Osimertinib Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Provencio, MD, Principal Investigator — Hospital Universitario Puerta de Hierro
Locations (31):
- Spain (31):
  - ICO Badalona, Badalona, Barcelona
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela, Galicia
  - Complejo Hospitalario Universitario A Coruña, A Coruña, La Coruña
  - Hospital Universitario Dr. Negrín, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Príncipe de Asturias, Alcalá de Henares, Madrid
  - Hospital Universitario de Getafe, Getafe, Madrid
  - Hospital Universitari Son Espases, Palma de Mallorca, Mallorca
  - Hospital Universitario Son Llàtzer, Palma de Mallorca, Mallorca
  - Complejo Hospitalario Universitario de Vigo, Vigo, Pontevedra
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Lluís Alcanyís, Xàtiva, Valencia
  - Hospital General de Albacete, Albacete
  - Hospital General Universitario Alicante, Alicante
  - Hospital de Sant Pau, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital Dr. Josep Trueta, Girona
  - Hospital Universitario de Guadalajara, Guadalajara
  - Complejo Hospitalario de Jaén, Jaén
  - Complejo Asistencial Universitario de León, León
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital General Universitario de Málaga, Málaga
  - Hospital Clínico de Salamanca, Salamanca
  - Hospital Virgen del Rocío, Seville
  - Hospital Virgen de la Salud, Toledo
  - Hospital Universitari i Politécnic La Fe, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Hospital Clínico Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Provencio M, Terrasa J, Garrido P, Campelo RG, Aparisi F, Diz P, Aguiar D, Garcia-Giron C, Hidalgo J, Aguado C, Gonzalez JG, Esteban E, Gomez-Aldavari L, Moran T, Juan O, Chara LE, Marti JL, Castro RL, Ortega AL, Moreno EM, Coves J, Sanchez Pena AM, Bosch-Barrera J, Gastaldo AS, Nunez NF, Del Barco E, Cobo M, Isla D, Majem M, Navarro F, Calvo V. Osimertinib in advanced EGFR-T790M mutation-positive non-small cell lung cancer patients treated within the Special Use Medication Program in Spain: OSIREX-Spanish Lung Cancer Group. BMC Cancer. 2021 Mar 6;21(1):230. doi: 10.1186/s12885-021-07922-5. PMID 33676426
- See also: Web page of the sponsor where users can find more information about Fundación GECP studies — http://www.gecp.org